CLINICAL TRIAL: NCT02221284
Title: Alogliptin (Nesina) Tablets Specified Drug-use Survey "Type 2 Diabetes Mellitus: Combination Therapy With Hypoglycemic Drug (Insulin Preparation or Rapid-acting Insulin Secretagogues, Etc)"
Brief Title: Alogliptin Tablets Specified Drug-use Survey "Type 2 Diabetic Patients Receiving Combination Therapy With a Hypoglycemic Agent (e.g., Insulin Preparations or Rapid-acting Insulin Secretagogues)"
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 121-016; JapicCTI-142609 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Results first posted 2019-07-19 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Pharmacological therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — alogliptin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Alogliptin: Alogliptin 25 milligram (mg), tablets, orally, once daily, up to 12 months, along with an insulin preparations, with a rapid-acting insulin secretagogue (Glinide), with a SGLT-2 inhibitor, or the other diabetic drugs within 3 months prior to the start of alogliptin treatment or during the alogliptin treatment period in routine medical care.
  Interventions: Drug: Alogliptin

INTERVENTIONS:
Drug: Alogliptin — Alogliptin tablets
  Other Names: Nesina Tablets

SUMMARY:
The purpose of this survey is to evaluate the safety and efficacy of long-term use of alogliptin tablets (Nesina Tablets) in type 2 diabetic patients who have had an inadequate response to hypoglycemic agents (e.g., insulin preparations or rapid-acting insulin secretagogues)* in addition to dietary/exercise therapy. Participants will receive alogliptin as part of routine medical care.

* Patients receiving these hypoglycemic agents (excluding α-glucosidase inhibitors, thiazolidines, sulfonylureas, and biguanides) were excluded from existing specified drug-use surveys for alogliptin tablets.

DETAILED DESCRIPTION:
This survey was designed to evaluate the safety and efficacy of long-term use of alogliptin tablets (Nesina Tablets) in type 2 diabetic patients who have had an inadequate response to hypoglycemic agents (e.g., insulin preparations or rapid-acting insulin secretagogues) in addition to dietary/exercise therapy. Participants will receive alogliptin as part of routine medical care.

For adults, 25 mg of alogliptin is usually administered orally once daily.

ELIGIBILITY:
Inclusion Criteria:

-Type 2 diabetic patients meeting the following criteria are included in this survey:

Patients who have had an inadequate response to the following medications/therapies:

• Use of one hypoglycemic agent such as insulin preparations and rapid-acting insulin secretagogues, excluding other types of hypoglycemic agents (e.g., α-glucosidase inhibitors, thiazolidines, sulfonylureas, and biguanides)*, in addition to dietary/exercise therapy

* For use of alogliptin tablets in combination with these agents, a specified drug-use survey is currently ongoing.

Exclusion Criteria:

-Type 2 diabetic patients who meet any of the following criteria are excluded from this survey: Patients with contraindications for alogliptin tablets

1. Those with severe ketosis, in a state of diabetic coma or precoma, or with type 1 diabetes mellitus [Quickly rectifying hyperglycemia with administration of intravenous fluid or insulin is essential in these patients; therefore, administration of alogliptin tablets is not appropriate.]
2. Those with severe infections, before or after surgery, or with serious trauma [Controlling blood glucose with an injection of insulin is desirable for these patients; therefore, administration of alogliptin tablets is not appropriate.]
3. Those with a history of hypersensitivity to any of the ingredients of alogliptin tablets

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type 2 diabetes mellitus
Sampling Method: Non-Probability Sample
Enrollment: 964 (Actual)
Dates: Start 2014-06-30 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (2):
- Japan (2):
  - Osaka
  - Tokyo

IPD SHARING:
Plan to Share IPD: No
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 196 investigative sites in Japan, from 30 June 2014 to 30 June 2017. Data reports overall population, since data not collected separately per arm as specified in protocol.
Pre-assignment Details: Enrolled participants had a diagnosis of type 2 diabetic mellitus and an inadequate response to hypoglycemic agents in addition to dietary/exercise therapy. Participants received interventions as part of routine medical care. Data reports overall population, since data not collected separately per arm as specified in protocol.
Groups:
- Overall Population: Alogliptin 25 milligram (mg), tablets, orally, once daily, up to 12 months, along with an insulin preparations, with a rapid-acting insulin secretagogue (Glinide), with a SGLT-2 inhibitor, or the other diabetic drugs within 3 months prior to the start of alogliptin treatment or during the alogliptin treatment period in routine medical care.
Period: Overall Study
Arm/Group | Overall Population
Started | 964
Completed | 903
Not Completed | 61
Not completed — Case Report Forms Uncollected | 56
Not completed — Protocol Deviation | 5

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set; The safety analysis set was defined as all participants who completed the study.
Groups:
- Alogliptin + Insulin: Alogliptin 25 mg, tablets, orally, once daily for up to 12 months, along with insulin preparation within 3 months prior to the start of alogliptin treatment or during the alogliptin treatment period. Participants received interventions as part of routine medical care.
- Alogliptin + Glinide: Alogliptin 25 mg, tablets, orally, once daily for up to 12 months, along with rapid-acting insulin secretagogue (Glinide) within 3 months prior to the start of alogliptin treatment or during the alogliptin treatment period. Participants received interventions as part of routine medical care.
- Alogliptin + SGLT-2 Inhibitor: Alogliptin 25 mg, tablets, orally, once daily for up to 12 months, along with SGLT-2 inhibitor within 3 months prior to the start of alogliptin treatment or during the alogliptin treatment period. Participants received interventions as part of routine medical care.
- Alogliptin + Other: Alogliptin 25 mg, tablets, orally, once daily for up to 12 months, along without insulin preparations, glinide, or SGLT-2 inhibitor within 3 months prior to the start of alogliptin treatment or during the alogliptin treatment period. Participants received interventions as part of routine medical care.
- Total: Total of all reporting groups
Arm/Group | Alogliptin + Insulin | Alogliptin + Glinide | Alogliptin + SGLT-2 Inhibitor | Alogliptin + Other | Total
Number analyzed (Participants) | 573 | 166 | 102 | 62 | 903
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.6 (12.27) | 67.9 (11.71) | 61.0 (13.72) | 61.2 (14.31) | 65.2 (12.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 257 | 67 | 35 | 26 | 385
  Male | 316 | 99 | 67 | 36 | 518
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  Japan | 573 | 166 | 102 | 62 | 903
Duration of Diagnosis of Type-2 Diabetes Mellitus (Years) [Mean (Standard Deviation); unit: Years] — Mean duration between start of study and first time of diagnosis of type 2 diabetes mellitus was reported. Population: The number analyzed is the number of participants with data available for analysis.
  Years
    number analyzed (Participants) | 417 | 120 | 34 | 50 | 621
    (all) | 14.24 (10.858) | 9.03 (9.058) | 6.57 (6.911) | 7.45 (6.831) | 12.26 (10.458)
Height [Mean (Standard Deviation); unit: Centimeters (cm)] — Population: The number analyzed is the number of participants with data available for analysis.
  Centimeters (cm)
    number analyzed (Participants) | 523 | 155 | 75 | 50 | 803
    (all) | 160.0 (9.70) | 160.2 (10.12) | 164.3 (9.38) | 162.4 (9.02) | 160.6 (9.78)
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] — Population: The number analyzed is the number of participants with data available for analysis.
  Kilograms (kg)
    number analyzed (Participants) | 516 | 146 | 101 | 49 | 812
    (all) | 62.57 (12.910) | 62.45 (13.141) | 72.37 (14.654) | 68.32 (14.248) | 64.11 (13.667)
BMI [Median (Standard Deviation); unit: kg/meter (m)^2] — Body Mass Index = weight (kg)/[height (m)^2] Population: The number analyzed is the number of participants with data available for analysis.
  kg/meter (m)^2
    number analyzed (Participants) | 488 | 140 | 75 | 46 | 749
    (all) | 24.40 (4.037) | 24.22 (3.515) | 26.71 (4.380) | 25.90 (4.312) | 24.69 (4.065)
Waist Circumference (Male) [Count of Participants; unit: Participants] — Population: This baseline characteristic was analyzed only in male participants.
  Participants
    < 85 cm: number analyzed (Participants) | 316 | 99 | 67 | 36 | 518
    < 85 cm | 15 | 12 | 2 | 1 | 30
    >= 85 cm: number analyzed (Participants) | 316 | 99 | 67 | 36 | 518
    >= 85 cm | 22 | 17 | 9 | 5 | 53
    Unknown: number analyzed (Participants) | 316 | 99 | 67 | 36 | 518
    Unknown | 279 | 70 | 56 | 30 | 435
Waist Circumference (Female) [Count of Participants; unit: Participants] — Population: This baseline characteristic was analyzed only in female participants.
  Participants
    < 90 cm: number analyzed (Participants) | 257 | 67 | 35 | 26 | 385
    < 90 cm | 25 | 13 | 2 | 1 | 41
    >= 90 cm: number analyzed (Participants) | 257 | 67 | 35 | 26 | 385
    >= 90 cm | 15 | 3 | 2 | 1 | 21
    Unknown: number analyzed (Participants) | 257 | 67 | 35 | 26 | 385
    Unknown | 217 | 51 | 31 | 24 | 323
Healthcare Category [Count of Participants; unit: Participants] — Participants were categorized as outpatient and inpatient.
  Participants
    Outpatient | 539 | 161 | 101 | 57 | 858
    Inpatient | 34 | 5 | 1 | 5 | 45
Medical Complications [Count of Participants; unit: Participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above.
  Participants
    Had No Medical Complications | 69 | 18 | 21 | 14 | 122
    Had Medical Complications | 504 | 148 | 81 | 48 | 781
Concomitant Diabetes Mellitus [Count of Participants; unit: Participants]
  Had No Concomitant Diabetes Mellitus | 324 | 123 | 65 | 44 | 556
  Had Concomitant Diabetes Mellitus | 249 | 43 | 37 | 18 | 347
Concomitant Hypertension [Count of Participants; unit: Participants]
  Had No Concomitant Hypertension | 247 | 63 | 41 | 26 | 377
  Had Concomitant Hypertension | 326 | 103 | 61 | 36 | 526
Concomitant Hyperlipidemia [Count of Participants; unit: Participants]
  Had No Concomitant Hyperlipidemia | 261 | 68 | 38 | 29 | 396
  Had Concomitant Hyperlipidemia | 312 | 98 | 64 | 33 | 507
Concomitant Hyperuricaemia [Count of Participants; unit: Participants]
  Had No Concomitant Hyperuricaemia | 522 | 145 | 93 | 60 | 820
  Had Concomitant Hyperuricaemia | 51 | 21 | 9 | 2 | 83
Concomitant Hepatic Disorder [Count of Participants; unit: Participants]
  Had No Concomitant Hepatic Disorder | 467 | 147 | 84 | 51 | 749
  Had Concomitant Hepatic Disorder | 106 | 19 | 18 | 11 | 154
Degree of Hepatic Dysfunction [Count of Participants; unit: Participants] — Severity was determined using aspartate aminotransferase (AST) or alanine transaminase (ALT) values at the start of treatment with alogliptin. For the assessment of severity, the following categories were used and higher grades of serum AST or ALT were adopted. Normal: <50 units per liter (U/L) Grade 1: >=50 to <100 U/L Grade 2: >=100 to <500 U/L Grade 3: >=500 U/L
  Participants
    Normal | 404 | 94 | 63 | 36 | 597
    Grade 1 | 25 | 7 | 5 | 4 | 41
    Grade 2 | 4 | 3 | 5 | 1 | 13
    Unknown | 140 | 62 | 29 | 21 | 252
Concomitant Renal Disorder [Count of Participants; unit: Participants]
  Had No Concomitant Renal Disorder | 412 | 139 | 73 | 49 | 673
  Had Concomitant Renal Disorder | 161 | 27 | 29 | 13 | 230
Degree of Renal Dysfunction (eGFR) [Count of Participants; unit: Participants] — Estimated glomerular filtration rate (eGFR) was calculated using variables of gender, age at the start of treatment, and serum creatinine values, and severity was determined based on the following categories. If the serum creatinine value or age at the start of treatment was not listed, the severity was reported as "unknown". Normal: >=90 milliliter per min (mL/min)/1.73^2, Mild: >=60 mL/min/1.73^2 to <90 mL/min/1.73^2, Moderate: >=30 mL/min/1.73^2 to <60 mL/min/1.73^2, Severe: <30 mL/min/1.73^2; eGFR= 194 * Cr^-1.094 * (age)^-0.287 (* 0.739 if female) where Cr is creatinine value.
  Participants
    Normal | 85 | 30 | 23 | 16 | 154
    Mild | 235 | 38 | 38 | 22 | 333
    Moderate | 118 | 28 | 18 | 4 | 168
    Severe | 12 | 1 | 0 | 0 | 13
    Normal or Mild | 320 | 68 | 61 | 38 | 487
    Moderate or Severe | 130 | 29 | 18 | 4 | 181
    Unknown | 123 | 69 | 23 | 20 | 235
Degree of Renal Dysfunction (Cr) [Count of Participants; unit: Participants] — Normal or Mild: =< 1.4 mg/dL (for male) or =< 1.2 mg/dL (for female), Moderate: >1.4 mg/dL to =< 2.4 mg/dL (for male) or >1.2 mg/dL to =< 2.0 mg/dL (for female), Severe: > 2.4 mg/dL (for male), > 2.0 mg/dL (for female). If the serum creatinine value (Cr) at the start of treatment was not listed, the severity was reported as "unknown".
  Participants
    Normal or Mild | 431 | 94 | 78 | 42 | 645
    Moderate | 17 | 3 | 1 | 0 | 21
    Severe | 2 | 0 | 0 | 0 | 2
    Moderate or Severe | 19 | 3 | 1 | 0 | 23
    Unknown | 123 | 69 | 23 | 20 | 235
Concomitant Cardiac Disease [Count of Participants; unit: Participants]
  Had No Concomitant Cardiac Disease | 467 | 154 | 96 | 54 | 771
  Had Concomitant Cardiac Disease | 106 | 12 | 6 | 8 | 132
Concomitant Heart Failure [Count of Participants; unit: Participants]
  Had No Concomitant Heart Failure | 546 | 166 | 101 | 61 | 874
  Had Concomitant Heart Failure | 27 | 0 | 1 | 1 | 29
New York Heart Association (NYHA) Heart Failure Classification [Count of Participants; unit: Participants] — NYHA functional classification ranges from Class I (participants with cardiac disease but without resulting limitations of physical activity), Class II (participants with cardiac disease resulting in slight limitation of physical activity), Class III (participants with cardiac disease resulting in marked limitation of physical activity), Class IV (participants with cardiac disease resulting in inability to carry on any physical activity without discomfort). Population: This baseline characteristic was analyzed only for participants who had complications of heart failure.
  Participants
    Class I: number analyzed (Participants) | 27 | 0 | 1 | 1 | 29
    Class I | 15 | 0 | 0 | 1 | 16
    Class II: number analyzed (Participants) | 27 | 0 | 1 | 1 | 29
    Class II | 9 | 0 | 1 | 0 | 10
    Unknown: number analyzed (Participants) | 27 | 0 | 1 | 1 | 29
    Unknown | 3 | 0 | 0 | 0 | 3
Concomitant Stroke-Related Disease [Count of Participants; unit: Participants]
  Had No Concomitant Stroke-Related Disease | 520 | 157 | 99 | 61 | 837
  Had Concomitant Stroke-Related Disease | 53 | 9 | 3 | 1 | 66
Concomitant Allergic Condition [Count of Participants; unit: Participants]
  Had No Concomitant Allergic Condition | 553 | 161 | 99 | 59 | 872
  Had Concomitant Allergic Condition | 20 | 5 | 3 | 3 | 31
Concomitant Malignant Tumor [Count of Participants; unit: Participants]
  Had No Concomitant Malignant Tumor | 548 | 160 | 102 | 59 | 869
  Had Concomitant Malignant Tumor | 25 | 6 | 0 | 3 | 34
Medical History [Count of Participants; unit: Participants] — Medical history defined as a disease or a health condition for each participant before start of the study. Medical history was classified as congenital anomalies, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, GI disorders, hepatic and biliary disorders, renal disease and other medical history. Other medical history included all medical history except for those mentioned above.
  Participants
    Had No Medical History | 411 | 123 | 95 | 47 | 676
    Had Medical History | 125 | 28 | 5 | 12 | 170
    Unknown | 37 | 15 | 2 | 3 | 57
Predisposition to Hypersensitivity [Count of Participants; unit: Participants] — The baseline characteristic was analyzed in participants who had a liability or tendency to suffer from hypersensitivity.
  Participants
    Had No Predisposition to Hypersensitivity | 508 | 141 | 98 | 56 | 803
    Had Predisposition to Hypersensitivity | 33 | 11 | 3 | 4 | 51
    Unknown | 32 | 14 | 1 | 2 | 49
Drinking Habits [Count of Participants; unit: Participants] — Participants who answered Yes or No for a question "Drink Alcohol Almost Every Day?" were reported.
  Participants
    Yes | 110 | 49 | 23 | 14 | 196
    No | 377 | 92 | 57 | 39 | 565
    Unknown | 86 | 25 | 22 | 9 | 142
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 289 | 65 | 43 | 25 | 422
  Current Smoker | 64 | 31 | 15 | 16 | 126
  Ex-Smoker | 103 | 45 | 19 | 10 | 177
  Unknown | 117 | 25 | 25 | 11 | 178
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percent] — Population: The number analyzed is the number of participants with data available for analysis.
  Percent
    number analyzed (Participants) | 559 | 160 | 96 | 61 | 876
    (all) | 8.44 (1.662) | 7.60 (1.051) | 7.66 (1.379) | 8.78 (2.053) | 8.21 (1.612)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Had One or More Adverse Reactions
Description: Adverse drug reactions are defined as adverse events (AEs) which are in the investigator's opinion of causal relationship to the study treatment. AEs are defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug.
Time Frame: Up to Month 12
Population: Safety Analysis Set; The safety analysis set was defined as all participants who completed the study.
Measure: Number; unit: Percentage of Participants
Arm/Group | Alogliptin + Insulin | Alogliptin + Glinide | Alogliptin + SGLT-2 Inhibitor | Alogliptin + Other
Number analyzed (Participants) | 573 | 166 | 102 | 62
Percentage of Participants | 5.41 | 1.20 | 0.98 | 0.00

2. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c)
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at final assessment point (up to Month 12) relative to baseline.
Time Frame: Baseline, and final assessment point (up to Month 12)
Population: Efficacy assessment population was defined as participants who completed study and had available efficacy data at baseline and post baseline. Efficacy analysis was planned to be assessed in Alogliptin + Insulin, Alogliptin + Glinide and Alogliptin + SGLT-2 inhibitor groups and data for Alogliptin + Other were not collected as specified in protocol.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Alogliptin + Insulin | Alogliptin + Glinide | Alogliptin + SGLT-2 Inhibitor
Number analyzed (Participants) | 546 | 158 | 96
Percent | -0.66 (1.622) | -0.49 (0.940) | -0.60 (1.102)

3. Secondary Outcome: Number of Participants Achieving Specified HbA1c Level (< 7.0% and <6.0%)
Description: The reported data were number of participants who achieved specified HbA1c Level (< 7.0% and <6.0%) during this study.
Time Frame: Baseline, and final assessment point (up to Month 12)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Alogliptin + Insulin | Alogliptin + Glinide | Alogliptin + SGLT-2 Inhibitor
Number analyzed (Participants) | 557 | 162 | 101
Participants
  HbA1c Level < 7.0% | 161 | 87 | 55
  HbA1c Level < 6.0% | 22 | 10 | 7

4. Secondary Outcome: Change From Baseline in Laboratory Test Values (Fasting Blood Glucose Level)
Description: The reported data were change from baseline in fasting blood glucose level.
Time Frame: Baseline, and final assessment point (up to Month 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Milligram (mg)/deciliter (dL)
Arm/Group | Alogliptin + Insulin | Alogliptin + Glinide | Alogliptin + SGLT-2 Inhibitor
Number analyzed (Participants) | 87 | 33 | 21
Milligram (mg)/deciliter (dL) | -16.4 (65.96) | -32.0 (42.00) | -18.7 (35.86)

5. Secondary Outcome: Change From Baseline in Laboratory Test Values (Fasting Insulin Level)
Description: The reported data were change from baseline in fasting insulin level.
Time Frame: Baseline, and final assessment point (up to Month 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Micro Units per Milliliter (μU/mL)
Arm/Group | Alogliptin + Insulin | Alogliptin + Glinide | Alogliptin + SGLT-2 Inhibitor
Number analyzed (Participants) | 5 | 10 | 1
Micro Units per Milliliter (μU/mL) | -3.08 (3.414) | 2.26 (4.948) | 0.40 (NA) — Standard Deviation was not calculated as only one participant was analyzed.

6. Secondary Outcome: Change From Baseline in Laboratory Test Values (Homeostasis Model Assessment Ratio [HOMA-R])
Description: The reported data were change from baseline in HOMA-R. HOMA-R measures insulin resistance, calculated by fasting insulin (μU/mL) multiplied by fasting glucose (mg/dL), and divided by a constant (405). A higher score indicates higher insulin resistance.
Time Frame: Baseline, and final assessment point (up to Month 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: HOMA-R Score
Arm/Group | Alogliptin + Insulin | Alogliptin + Glinide | Alogliptin + SGLT-2 Inhibitor
Number analyzed (Participants) | 5 | 10 | 1
HOMA-R Score | -2.58 (2.170) | -0.25 (2.094) | 0.00 (NA) — Standard Deviation was not calculated as only one participant was analyzed.

7. Secondary Outcome: Change From Baseline in Laboratory Test Values (Homeostasis Model Assessment of Beta-cell Function [HOMA-β])
Description: The reported data were change from baseline in HOMA-β. HOMA-β measures as following; HOMA-β = fasting insulin (μU/mL) ×360/{fasting glucose (mg/dL) - 63}.
Time Frame: Baseline, and final assessment point (up to Month 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of beta cell function
Arm/Group | Alogliptin + Insulin | Alogliptin + Glinide | Alogliptin + SGLT-2 Inhibitor
Number analyzed (Participants) | 5 | 10 | 1
Percentage of beta cell function | 12.32 (17.286) | 33.38 (19.851) | 15.40 (NA) — Standard Deviation was not calculated as only one participant was analyzed.

ADVERSE EVENTS:
Time Frame: Up to Month 12
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Only adverse drug reactions (ADRs) were collected and reported on safety results sections here. ADRs are adverse events (AEs) which are in the investigator's opinion of causal relationship to the study treatment.
Groups:
- Alogliptin + SGLT-2 Inhibit: Alogliptin 25 mg, tablets, orally, once daily for up to 12 months, along with SGLT-2 inhibitor within 3 months prior to the start of alogliptin treatment or during the alogliptin treatment period. Participants received interventions as part of routine medical care.
Arm/Group | Alogliptin + Insulin | Alogliptin + Glinide | Alogliptin + SGLT-2 Inhibit | Alogliptin + Other
All-Cause Mortality (participants affected / at risk) | 3/573 | 0/166 | 0/102 | 0/62
Serious Adverse Events (participants affected / at risk) | 3/573 | 0/166 | 0/102 | 0/62
Other Adverse Events (participants affected / at risk) | 10/573 | 2/166 | 0/102 | 0/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin + Insulin (N=573) | Alogliptin + Glinide (N=166) | Alogliptin + SGLT-2 Inhibit (N=102) | Alogliptin + Other (N=62)
Cardiac failure acut (Cardiac disorders) | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Death (General disorders) | 1 | 0 | 0 | 0 — The reasons of events are not determined because assessment findings were insufficient to specify the reason.
OTHER ADVERSE EVENTS (reported when occurring in more than 1.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin + Insulin (N=573) | Alogliptin + Glinide (N=166) | Alogliptin + SGLT-2 Inhibit (N=102) | Alogliptin + Other (N=62)
Hypoglycaemia (Metabolism and nutrition disorders) | 7 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2017-06-02): https://cdn.clinicaltrials.gov/large-docs/84/NCT02221284/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-11): https://cdn.clinicaltrials.gov/large-docs/84/NCT02221284/SAP_001.pdf